CLINICAL TRIAL: NCT03996967
Title: Diagnostic and Prognostic Biomarkers for Childhood Bacterial Pneumonia in Sub-Saharan Africa
Brief Title: Diagnostic and Prognostic Biomarkers for Childhood Bacterial Pneumonia
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Medical Research Council Unit, The Gambia, LSTMH (Unknown); Laboratory of Transnational Immunology, UMC Utrecht (Unknown)
Responsible Party: Sponsor
Other Study IDs: H-38462; R21AI140258-01 (NIH)
Record Dates: First submitted 2019-06-20; First posted 2019-06-25 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Pneumonia, Bacterial; Viral Infection; Clinical Pneumonia; Plasmodium Falciparum Malaria; Malaria; Infections, Respiratory
Keywords: Biosignature proteins; Luminex®-based immunoassays; Point-of-care test; Children; Sub-Saharan Africa; Diagnostic Biomarkers; Prognostic Biomarkers; Mediators of Inflammation
MeSH Terms: conditions — Pneumonia, Bacterial; Virus Diseases; Malaria, Falciparum; Malaria; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood will be collected from 900 children hospitalized with pneumonia for the multiplex bead-based immunoassay and for tests that will be part of standard of care, including full blood cell count, bacterial blood culture, rapid malaria test and/or blood smear slide for malaria diagnosis. Also as part of standard of care in PVS, a nasopharyngeal swab will be collected, and analyzed in this study for viral PCR. Venous blood for the multiplex bead-based immunoassay will also be collected from 20 healthy controls to evaluate the precision of the biomarkers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BA Group: The bacterial group: Patients will be assorted to this group if he/she has a bacterial pathogen culture of fluid from a normally sterile site (e.g. blood, pleural fluid)
- VI Group: The viral group: Patients will be assigned to this group if they have negative bacteria microbiological tests, negative malaria blood slides, X-rays without "endpoint pneumonia", no evidence of fungal infection, and positive PCR for a viral pathogen from nasopharyngeal swabs.
- MA Group: The malarial group: Patients will be assigned to this group if they have normal X-rays, no bacterial infection and >0 asexual P. falciparum parasites if they are aged < 1 year, or > 2,500 asexual parasites/µl of blood if they are aged > 1 year

SUMMARY:
Clinical pneumonia is a leading cause of pediatric hospitalization. The etiology is generally bacterial or viral. Prompt and optimal treatment of pneumonia is critical to reduce mortality. However, adequate pneumonia management is hampered by: a) the lack of a diagnostic tool that can be used at point-of-care (POC) and promptly and accurately allow the diagnosis of bacterial disease and b) lack of a prognostic POC test to help triage children in need of intensive assistance. Antibiotic therapy is frequently overprescribed as a result of suspected bacterial infections resulting in development of antibiotic resistance. Conversely, in malaria-endemic areas, antibiotics may also be "underprescribed" and children with bacterial pneumonia sent home without antibiotic therapy, when the clinical pneumonia is mistakenly attributed to a co-existing malaria infection.

The investigators previously identified combinations of protein with 96% sensitivity and 86% specificity for detecting bacterial disease in Mozambican children with clinical pneumonia. The investigators' prior work showed that it is possible to identify biosignatures for diagnosis and prognosis using few proteins. Recently, other authors also identified different accurate biosignatures (e.g., IP-10, TRAIL and CRP).

In this study, the investigators propose to validate and improve upon previous biosignatures by testing prior combinations and seeking novel combinations of markers in 900 pediatric inpatients aged 2 months to 5 years with clinical pneumonia in The Gambia. The investigators will also use alternative case criteria and seek diagnostic and prognostic combination of markers. This study will be conducted in Basse, rural Gambia, in two hospitals associated with the Medical Research Council Unity The Gambia (MRCG). Approximately 900 pediatric patients with clinical pneumonia aged 2 months to 5 years of age will be enrolled. Patients will undergo standard of care test and will have blood proteins measured through Luminex®-based immunoassays.

Results of this study may ultimately support future development of an accurate point-of-care test for bacterial disease to guide clinicians in choices of treatment and to assist in the prioritization of intensive care in resource-limited settings.

ELIGIBILITY:
Inclusion criteria Clinical Pneumonia Patients

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Pediatric patients aged between 2 months and 5 years presenting at the screening sites with respiratory symptoms, i.e. cough or difficulty breathing AND
* One of the following: Increased respiratory rate for age OR indrawing OR SaO2 < 93% OR grunting OR MUAC < 11.5 if child is greater or equal than 6 months of age OR visible wasting AND
* Referred to clinician review for probable admission

Definition of increased respiratory rate (rr) for age based on the WHO criteria: respiratory rate (rr) > > 50 for 2-11 month old; rr > 40 for 1-5 years old.

Inclusion criteria Healthy Controls

* No symptoms or signs of any disease
* No malaria infection as detected by microscopy or RDT
* No history of clinical pneumonia or hospital admission

Exclusion criteria Clinical Pneumonia Patients

An individual who meets any of the following criteria will be excluded from participation in this study:

* Suspected tuberculosis based on history of cough lasting > 2 weeks
* Hospital admission in the previous 2 weeks.
* Children that show any evidence of other conditions that could be worsened by blood collection will be further excluded from this study.

Exclusion criteria Healthy Controls

• Having received a vaccine within the prior 4 weeks

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will be enrolling children 2 month-5 years of age who seek treatment for clinical pneumonia at two hospitals in rural Gambia: Basse and Bansang hospitals
Sampling Method: Non-Probability Sample
Enrollment: 837 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Definitive diagnosis of an invasive bacterial disease (versus viral and malarial infection) | At admission
  A patient will be assigned to the bacterial (BA) group if he/she has a bacterial pathogen culture of fluid from a normally sterile site (e.g. blood, pleural fluid). Patients will be assigned to the viral (VI) group if they have negative bacteria microbiological tests, negative malaria blood slides, X-ray without "endpoint pneumonia" (consolidation or pleural effusion50), no evidence of fungal infection, and positive PCR for a viral pathogen from nasopharyngeal swabs. Patients will be assigned to the malarial (MA) group if they have normal X-ray (with neither infiltrates nor endpoint pneumonia), no bacterial infection and > 0 asexual P. falciparum parasites if they are aged < 1 year, or > 2,500 asexual parasites/µl of blood if they are aged > 1 year. Patients who are admitted with viral infections but who develop bacterial pneumonia during hospitalization will be excluded from VI
Poor prognosis of clinical pneumonia | 30 days from admission
  Patients will be categorized in the following three groups based on a review of clinical records: a) children who die during or within the first 30 days from admission (all children that meet this criteria), b) children with prolonged hospital stay or who need to have antibiotic therapy changed within 48 hours of admission or who were re-admitted within 30 days from the first admission; and c) children discharged well within 3 days of admission and without the need for a change in antibiotic therapy after admission.

SECONDARY OUTCOMES:
Probable bacterial pneumonia (versus viral pneumonia or severe malaria) | At admission
  Based on the review of data by an expert panel, patients will be assigned to either: a) the probable bacterial group (BA) or the b) non bacterial group. Data to be reviewed by the panel will include chest X-ray, complete blood cell counts, other laboratory results, the clinical course during admission and following discharge. Children will be assigned to the non bacterial group (i.e, VI or MA) if they have X-ray without endpoint pneumonia, pleural effusion or infiltrates, do not have bacterial infection as per the algorithm for definitive diagnosis and are not classified as bacterial infection by the expert panel.
Oxygen saturation curve | Within the first 5 days of admission
  Area under the first five days of the oxygen saturation curve. Oxygen saturation will be recorded daily in the morning in a follow-up form
Need to switch antibiotic therapy | Within the first 3 days of admission
  All patients will be classified as either needing or not needing to switch within the first three days of hospitalization their antibiotic therapy prescribed at admission based on a follow-up form
Duration of hospital admission | Within 3 days of hospital discharge
  The total length of hospital admission will be calculated in days for each patient based on the difference between the dates of discharge and admission.
Time to start feeding well | Within the first 5 days of admission
  Time to feed well will be defined based on the child examination in the morning within the first 5 days of follow-up that will be recorded in a follow-up form

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa Valim, MD ScD, Principal Investigator — Boston University; Patricia Hibberd, MD PhD, Principal Investigator — Boston University
Locations (3):
- Boston University School of Public Health, Boston, Massachusetts, United States
- Laboratory of Transnational Immunology, UMC Utrecht, Utrecht, Netherlands
- Basse Field Station, Medical Research Council Gambia Unit, Basse Santa Su, URR, The Gambia

IPD SHARING:
Plan to Share IPD: No